CLINICAL TRIAL: NCT02177513
Title: Effects of Cannabis Administration Routes on Human Performance and Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 999914135; 14-DA-N135
Record Dates: First submitted 2014-06-24; First posted 2014-06-27 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2016-04-27

CONDITIONS: Cannabis Use
Keywords: Cannabis; Pharmacodynamics; Marijuana; Cannabinoids; Vaporized
MeSH Terms: conditions — Marijuana Abuse | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (5):
- 1 (Active Comparator)
  Interventions: Drug: Placebo + Smoked Cannabis
- 2 (Active Comparator)
  Interventions: Drug: Placebo + Inhaled Cannabis
- 3 (Active Comparator)
  Interventions: Drug: Oral Cannabis + Placebo
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo + Placebo
- 5 (Active Comparator)
  Interventions: Drug: 6.9% cannabis oral

INTERVENTIONS:
Drug: Placebo + Placebo — Participants will consume a brownie containing the equivalent of one placebo (0.001% THC) cigarette followed by smoking or inhaling (after vaporization) the equivalent of one placebo (0.001% THC) cigarette.
  Arms: 4
Drug: Oral Cannabis + Placebo — Participants will consume a brownie containing the equivalent of one active (6.9% THC) cannabis cigarette followed by either smoking or inhaling (after vaporization) the equivalent of one placebo (0.001% THC) cigarette.
  Arms: 3
Drug: Placebo + Inhaled Cannabis — Participants will consume a brownie containing the equivalent of one placebo (0.001% THC) cigarette
  Arms: 2
Drug: Placebo + Smoked Cannabis — Participants will consume a brownie containing the equivalent of one placebo (0.001% THC) cigarette followed by smoking the equivalent of one active (6.9% THC) cigarette.
  Arms: 1
Drug: 6.9% cannabis oral — Participants will consume a brownie containing the equivalent of one active (6.91% THC) cannabis cigarette.
  Arms: 5

SUMMARY:
Background:

- Marijuana (cannabis) is an illegal drug. Researchers want to study people s reactions, attention, and behavior after they take marijuana in different ways. They want to learn better ways to detect drugs in a person s body They also want to know how long marijuana can be found in blood, urine, saliva, and breath.

Objectives:

- To learn how people respond to delta-9-tetrahydrocannabinol (THC, a marijuana component) and how their bodies handle it after it is given in different ways.

Eligibility:

- Adults age 18 50 who use marijuana.

Design:

* Participants are screened under another NIDA protocol.
* This study involves up to 6 visits to NIDA.
* At the first visit, participants will practice the tasks and tests they will do at their dosing sessions. They will learn how to give breath and saliva samples.
* Dosing sessions 1 4 will last 3 5 days each. All participants will be admitted to a research clinic the night before these sessions. Some participants can stay at the clinic and some must go home between sessions.
* At each session, participants will eat a brownie with placebo or marijuana. Then they will smoke a placebo or marijuana cigarette. Some will inhale placebo or marijuana after it is vaporized.
* Throughout the sessions:
* Participants will give urine, saliva, and breath samples. Their blood will be taken with a tube in a vein and finger pricks. Their vital signs will be checked.
* Participants will answer questionnaires and take thinking tests. They will also take tests that assess eye movement, balance, and time estimation.
* Participants may have a 5th dosing session. They will eat a marijuana brownie and have the above tests and samples.

DETAILED DESCRIPTION:
Objectives

Cannabinoids are most commonly administered via smoking. Oral consumption in medications, teas, oils, or food also is widely utilized. Additionally, cannabis vaporization followed by inhalation for medical and illicit administration is common. Differences in cannabis pharmacodynamics and pharmacokinetics between these three administration routes and in occasional and frequent cannabis smokers are not thoroughly characterized. This study evaluates cannabis pharmacodynamics and pharmacokinetics in occasional and frequent smokers after smoked, vaporized, and oral cannabis administration.

<TAB>

Study Population

Up to 80 healthy cannabis smokers, aged 18-50, without a history of adverse reactions to cannabis will be recruited. For dosing sessions 1-4, ten occasional smokers (smoking frequency greater than or equal to 2 times/month but <3 times/week) and ten frequent smokers (smoking frequency generally greater than or equal to 5times/week) are required. For the optional 5th session, 8-20 participants (regardless of smoking history) are required.

<TAB>

Study Design

Occasional and frequent cannabis smokers are recruited to participate. Prior to dosing sessions, there is a training visit for all study procedures. Sessions 1-4 are 3 and 4 days each for occasional and frequent cannabis smokers, respectively, and the study design is double blind, double dummy, randomized, crossover, and placebo-controlled. In each session, participants will consume a placebo or active oral (baked in a brownie) cannabis (6.9% 9-tetrahydrocannabinol [THC]) dose followed by either placebo or active smoked or vaporized cannabis. Only one active dose will be administered in each dosing session. Whole blood, oral fluid, urine, dried blood spots, and breath are collected throughout all sessions. Due to the large THC body burden stored in the tissues, we will collect biological specimens for a longer period in frequent cannabis smokers than for occasional cannabis smokers. An optional 5th dosing session will be offered in which participants receive a single oral cannabis dose for pharmacokinetic monitoring. The placebo cannabis plant material has a low THC concentration. As we are expecting that the active brownie dose might result in low THC oral fluid contamination, it is necessary to have an active brownie THC dose that is not followed by placebo vaporizer or smoked cannabis. Occasional smokers may stay or be discharged between sessions, including between the 4th and optional 5th dosing session, but dosing must not exceed self-reported intake frequency. Frequent smokers must be discharged for at least 72 h between dosing sessions 1-4, and must stay on the unit at the end of session 4 for session 5 if they choose to participate. The difference between requirements for occasional and frequent smokers to participate in the optional 5th dose is due to the potential confound of low THC concentrations in frequent smokers that might not permit the detection of low THC concentrations after consumption of a low oral THC dose. Occasional cannabis smokers will reside on the closed research unit for approximately 72 h for dosing sessions 1-4, and for approximately 66 h for dosing session 5. Frequent cannabis smokers will reside on the closed research unit for approximately 90 h for dosing sessions 1-3 (and 4 if not participating in optional session 5). If a frequent smoker chooses to participate in dosing session 5, they will remain on the unit for approximately 162 h for sessions 4 and 5. Participants will complete a battery of subjective, objective, and neurocognitive tests before and after dosing. Subjective effects are assessed with visual analog scales. Objective measurements include physiological measurements, expired carbon monoxide, reddening of the conjunctivae and tests measuring psychomotor skills and cognitive functions.

<TAB>

Outcome Parameters

Primary outcome measures include subjective and objective assessments, performance on neurocognitive tasks, and cannabinoid concentrations in whole blood, oral fluid, urine, dried blood spots, and breath. Correlations between cannabinoid concentrations in whole blood, dried blood spots, oral fluid, and breath will be investigated, the Oral Fluid Working Group for the Partnership for Clean Competition oral fluid screening algorithm will be evaluated, and the pharmacokinetic profiles of alternative cannabinoids will be characterized. Secondary investigations include comparing cannabinoid stability in dried blood spots and whole blood, evaluating the World Anti-Doping Agency urine 11-nor-9-carboxy-THC decision limit, characterizing the performance of the Alere DDS2 on-site oral fluid screening device, and evaluating effects of acute cannabis administration on leptin and other appetitive peptides.<TAB>

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. 18 to 50 years of age;
  2. Cannabis consumption with a minimum frequency of at least twice per month during the three months prior to the study and average frequency of cannabis smoking of less than three times per week (occasional cannabis smoker) in the past 3 months or at least an average of five times per week (frequent cannabis smoker) in the past 3 months;
  3. A positive urine cannabinoid screen if in the frequent cannabis smoker group;
  4. Peripheral veins suitable for repeated venipuncture and/or placement of an intravenous catheter, as assessed by a physician s assistant, nurse, or physician;
  5. Blood pressure (BP) and heart rate (HR) at or below the following values while sitting after five min rest: systolic BP (SBP) 140 mm Hg, diastolic BP (DBP) 90 mm Hg, heart rate (HR) 100 bpm;
  6. ECG and three-minute rhythm strip without clinically relevant abnormalities;
  7. Women with reproductive potential must use a medically acceptable form of contraception for the duration of the study. Medically acceptable forms of contraception include: oral contraceptive, intrauterine device (IUD), depot hormonal preparation (ring, injection implant), or a barrier method of contraception such as a diaphragm, sponge with spermicide, or a condom. Abstinence is an alternative lifestyle and subjects practicing abstinence may be included in the study.
  8. Must be able to safely suspend use of CNS depressant, anticholinergic, and/or sympathomimetic medications before study dosing. Length of medication suspension will be equal to 3 half-lives of the medication in use.

EXCLUSION CRITERIA:

1. Current physical dependence on any drug other than cannabis, caffeine, or nicotine;
2. Currently using cannabis for medical purposes under the explicit recommendation of a physician providing medical care;
3. History or presence of any clinically significant illness, as detected by history, physical examination, and/or laboratory tests , that might put the subject at increased risk of adverse events such as history of psychotic disorder, clinically significant mood and/or anxiety disorder, diabetes, liver, renal or cardiovascular disease;
4. Liver enzymes greater than or equal to 2 times upper normal limit and/or clinical signs/symptoms consistent with liver disease including but not limited to nausea, vomiting, jaundice, itching, abdominal pain, and swelling;
5. History of clinically significant adverse events associated with cannabis intoxication such as severe anxiety and panic, paranoia and psychosis, sustained tachycardia, or severe hypotension;
6. Donation of more than 450 mL blood within 8 weeks of study treatment phase;
7. Hemoglobin less than 12.0 g/dL and/or clinical signs/symptoms consistent with anemia including but not limited to fatigue, tachycardia, shortness of breath, and dizziness;
8. If female, pregnant or nursing;
9. Currently interested in or participating in drug abuse treatment, or participated in drug abuse treatment within 90 days preceding study enrollment;
10. History of food allergy or sensitivity to gluten, dairy, egg, soy, and/or chocolate.
11. Any form of color blindness

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2014-06-14; Primary Completion 2016-04-27 (Actual); Study Completion 2016-04-27 (Actual)

PRIMARY OUTCOMES:
Cannabis' pharmacodynamic effects | Multiple times daily
Cannabis' pharmacokinetic profiles | Multiple times daily
Pharmacokinetic/Dynamic Modelling | Once
Cannabis oral fluid cutoff evaluation | Once

SECONDARY OUTCOMES:
Cannabinoid stability in dried blood | Multiple times
Pharmacokinetic/Dynamic Modelling | Multiple times
Cannabinoid stability in oral fluid | Multiple times
Cannabis' effects on appetitive peptides | Multiple times daily
Cannabis urine cutoff evaluation | Once
Compare on-site oral fluid devices | Once

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn Huestis, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

REFERENCES:
- [Background] Vega WA, Aguilar-Gaxiola S, Andrade L, Bijl R, Borges G, Caraveo-Anduaga JJ, DeWit DJ, Heeringa SG, Kessler RC, Kolody B, Merikangas KR, Molnar BE, Walters EE, Warner LA, Wittchen HU. Prevalence and age of onset for drug use in seven international sites: results from the international consortium of psychiatric epidemiology. Drug Alcohol Depend. 2002 Dec 1;68(3):285-97. doi: 10.1016/s0376-8716(02)00224-7. PMID 12393223
- [Background] Huestis MA. Pharmacokinetics and metabolism of the plant cannabinoids, delta9-tetrahydrocannabinol, cannabidiol and cannabinol. Handb Exp Pharmacol. 2005;(168):657-90. doi: 10.1007/3-540-26573-2_23. PMID 16596792
- [Background] Grotenhermen F. Pharmacokinetics and pharmacodynamics of cannabinoids. Clin Pharmacokinet. 2003;42(4):327-60. doi: 10.2165/00003088-200342040-00003. PMID 12648025
- [Derived] Newmeyer MN, Swortwood MJ, Andersson M, Abulseoud OA, Scheidweiler KB, Huestis MA. Cannabis Edibles: Blood and Oral Fluid Cannabinoid Pharmacokinetics and Evaluation of Oral Fluid Screening Devices for Predicting Delta9-Tetrahydrocannabinol in Blood and Oral Fluid following Cannabis Brownie Administration. Clin Chem. 2017 Mar;63(3):647-662. doi: 10.1373/clinchem.2016.265371. Epub 2017 Feb 10. PMID 28188235
- [Derived] Newmeyer MN, Swortwood MJ, Taylor ME, Abulseoud OA, Woodward TH, Huestis MA. Evaluation of divided attention psychophysical task performance and effects on pupil sizes following smoked, vaporized and oral cannabis administration. J Appl Toxicol. 2017 Aug;37(8):922-932. doi: 10.1002/jat.3440. Epub 2017 Jan 31. PMID 28138971
- [Derived] Newmeyer MN, Swortwood MJ, Barnes AJ, Abulseoud OA, Scheidweiler KB, Huestis MA. Free and Glucuronide Whole Blood Cannabinoids' Pharmacokinetics after Controlled Smoked, Vaporized, and Oral Cannabis Administration in Frequent and Occasional Cannabis Users: Identification of Recent Cannabis Intake. Clin Chem. 2016 Dec;62(12):1579-1592. doi: 10.1373/clinchem.2016.263475. Epub 2016 Oct 10. PMID 27899456